CLINICAL TRIAL: NCT05535543
Title: Assessment of the Effects of Prone Positioning Among ARDS Patients on Ventilation Homogenization by the Phase Iii Slope of the Volumetric Capnography
Brief Title: Change in the Phase III Slope of the Volumetric Capnography by Prone Positioning in Acute Respiratory Distress Syndrome
Status: Recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Olcay Dilken, MD, Istanbul University - Cerrahpasa
Other Study IDs: 05072022-3605
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Acute Respiratory Distress Syndrome; Ventilation Perfusion Mismatch; Respiratory Failure
Keywords: Acute Respiratory Distress Syndrome; Volumetric Capnography; phase iii slope; prone
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency | interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Baseline slope of phase iii: Severe ARDS patients who are intubated and mechanically ventilated and will undergo prone positioning
  Interventions: Procedure: Prone Positioning

INTERVENTIONS:
Procedure: Prone Positioning — Patients will be turned to prone position and they will be left in prone position for a duration of at least 16 hours to a maximum of 24 hours. This duration is recommended by the ARDS guidelines.

SUMMARY:
This study evaluates the effects of prone positioning on homogenization of ventilation.

DETAILED DESCRIPTION:
After initiation of mechanical ventilation and assessing the eligibility of the patient, informed consent will be taken from the closest kin. If eligible, following steps will be performed which are part of standard ARDS patient care.

1. Low-flow Pressure Volume curve and assessment of airway opening pressure
2. Calculation of recruitment to inflation ratio
3. Optimizing Positive End-Expiratory Pressure

Afterwards, phase III slope of the patient will be recorded at four timepoints:

Supine 1 (immediately before turning to prone position) Prone 1 (immediately after prone position) Prone 2 (at the end of the 16-24 hour prone cycle) Supine 2 (immediately after turning to supine position)

ELIGIBILITY:
Inclusion Criteria:

* ARDS criteria met
* intubated and mechanically ventilated as a result of respiratory failure
* PaO2/FiO2 <200

Exclusion Criteria:

* age older than 18
* Chronic pulmonary disease, pneumothoraces, intraabdominal hypertension (> 12 mmHg), pregnancy, not expected to survive >24 hours, hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult mixed critical care patients
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in phase iii slope of the volumetric capnograph | 16 to 24 hours (according to time spent in the prone position)
  phase iii slope is associated with the ventilation homogeneity
correlation of the phase iii slope with the recruitment to inflation ratio | 16 to 24 hours (according to time spent in the prone position)
  recruitment to inflation ratio is a simple bedside tool that indicates a higher possible recruitable lung with higher applied Positive End-Expiratory Pressure

SECONDARY OUTCOMES:
correlation of the phase iii slope with the Partial pressure of the arterial oxygen/ Fraction of inspired O2 concentration (PaO2/FiO2) ratio | 16 to 24 hours (according to time spent in the prone position)
  PaO2/FiO2 is markedly reduced in ARDS patients as a consequence of aeration loss

CONTACTS AND LOCATIONS:
Overall Officials: Olcay Dilken, MD, Principal Investigator — Hamidiye Etfal Hospital
Locations (1):
- Hamidiye Etfal Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No